CLINICAL TRIAL: NCT01768624
Title: Patient Information About Options for Treatment (PINOT) Follow up Study: Answering Important Questions in Home Dialysis and Conservative Care.
Brief Title: PINOT Follow-up Study in End-stage Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Sydney South West Area Health Service (Other Government); South West Sydney Local Health District (Other); Kidney Health Australia (Unknown)
Responsible Party: Sponsor
Other Study IDs: RM-1/12
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; dialysis; pre dialysis education; transplantation; conservative care
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dialysis; Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stage 5 chronic kidney disease: Patients receiving home hemodialysis Patients receiving home peritoneal dialysis Patients receiving center-based hemodialysis Patients who had a pre-emptive kidney transplant Patients who planned for renal conservative care
  Interventions: Procedure: dialysis, kidney transplant

INTERVENTIONS:
Procedure: dialysis, kidney transplant

SUMMARY:
The primary aims of the Patient INformation about Options for Treatment (PINOT) Follow-up Study are to determine the proportions of patients, identified in the 2009 PINOT cohort that:

(i)Made the transition to home dialysis, after an initial start on center-based dialysis.

(ii)Commenced dialysis, or a time-limited trial of dialysis within 3 years, after confirmed plans for conservative care.

The hypotheses to be tested in the PINOT follow-up study are:

1. 50% of stage 5 chronic kidney disease patients who plan for home dialysis do not commence home dialysis within 3 years, and instead remain on centre-based haemodialysis; and,
2. less than 15% of stage 5 chronic kidney disease patients who plan for conservative care commence dialysis within 3 years.

DETAILED DESCRIPTION:
The secondary aims of the follow-up study include:

(i) To assess the primary reasons patients did not transition to home dialysis, in the planned home dialysis group.

(ii)To compare 3 and 5 year survival rates among patients who commenced conservative care and patients who commenced renal replacement therapy.

(iii) To assess the types of dialysis utilisation over a 5 year time period among the total cohort of patients.

(iv)To determine how renal palliative care services were engaged for conservative care patients, and document the patient's place of death (i.e. hospital, hospice, home with community palliative care).

ELIGIBILITY:
Inclusion Criteria:

* Adults and children with end stage kidney disease (eGFR <15 ml/min) who commenced renal replacement therapy or conservative care in Australia between July and September 2009

Exclusion Criteria:

* Patients returning to dialysis after a failed transplant,
* Patients with acute renal failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with chronic kidney disease attending renal treatment centres in Australian public hospitals and private practices
Sampling Method: Non-Probability Sample
Enrollment: 721 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who make the transition to home dialysis, after an initial start on center-based hemodialysis. | 5 years

SECONDARY OUTCOMES:
The proportion of patients who commence dialysis, or have a time-limited trial of dialysis within 3 and 5 years, after a confirmed plan for conservative care. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rachael L Morton, PhD, Principal Investigator — University of Sydney
Locations (2):
- University of Sydney, Sydney, New South Wales, Australia
- University of Oxford, Headington, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Morton RL, Howard K, Webster AC, Snelling P. Patient INformation about Options for Treatment (PINOT): a prospective national study of information given to incident CKD Stage 5 patients. Nephrol Dial Transplant. 2011 Apr;26(4):1266-74. doi: 10.1093/ndt/gfq555. Epub 2010 Sep 6. PMID 20819955
- [Background] Morton RL, Turner RM, Howard K, Snelling P, Webster AC. Patients who plan for conservative care rather than dialysis: a national observational study in Australia. Am J Kidney Dis. 2012 Mar;59(3):419-27. doi: 10.1053/j.ajkd.2011.08.024. Epub 2011 Oct 20. PMID 22014401
- [Result] Morton RL, Webster AC, McGeechan K, Howard K, Murtagh FEM, Gray NA, Kerr PG, Germain MJ, Snelling P. Conservative Management and End-of-Life Care in an Australian Cohort with ESRD. Clin J Am Soc Nephrol. 2016 Dec 7;11(12):2195-2203. doi: 10.2215/CJN.11861115. Epub 2016 Oct 3. PMID 27697783